CLINICAL TRIAL: NCT05798429
Title: The Effect of Compassion Training on the Compassion Competencies and Ethical Sensitivities of Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aliye Yıldırım (Other)
Responsible Party: Sponsor-Investigator, Aliye Yıldırım, Nurse, Suleyman Demirel University
Organization: Suleyman Demirel University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Compassion in nursing
Record Dates: First submitted 2023-02-04; First posted 2023-04-04 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Compassion
Keywords: Nursing Students; compassion; Compassion Competence; Moral Sensitivity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental)
  Interventions: Other: compassion education
- control group (No Intervention)

INTERVENTIONS:
Other: compassion education — 6 weeks of compassion training
  Arms: experimental group

SUMMARY:
The aim of this thesis study is to determine the effect of compassion education on compassion adequacy and moral sensitivity in nursing students. The sample of the descriptive study consists of the first year nursing students studying at Süleyman Demirel University in the 2022-2023 academic year. The research will be carried out between October 2022 and September 2023. Research data will be collected from nursing students who volunteered to participate in the research by using the Personal Information Form, which includes the demographic characteristics of the students, the Compassion Adequacy Scale and the Modified Moral Sensitivity Scale for Nursing Students.

DETAILED DESCRIPTION:
Values have an important place in the nursing profession. In this context, it is necessary to know the concept of compassion, which is among the values of health care.

Since the concept of Compassion-Compassion takes place in many disciplines, it has many definitions. According to the Turkish Language Association, it is defined as 'the feeling of sadness and pity for the bad situation that a person or another living thing encounters' (TDK). In the Dictionary of Bioethics Terms, it is defined as "an emotion directed towards a person or group (sometimes other than human beings) in a difficult or worse situation" .

When compassion is considered in the nursing profession, it is seen as an ethical obligation. The ethical codes and declarations of the American Nurses Association and the International Council of Nurses are also based on compassion .

While talking about care in Roach, he suggested that the concept of compassion is one of the characteristics that a caregiver should have . Cummings and Bennett defined the features required for the formation of a care culture with the concept of 6 Cs and emphasized that compassion is important here .

Compassion can be learned and developed from the environment and conditions. The purpose of education is to provide individuals with certain behaviors. Explaining compassion education to students not only increases compassion towards other individuals, but also allows them to have positive emotions, integrating the coping methods they have gained into their own lives, increasing their feelings of compassion towards themselves.

The concept of compassion adequacy was defined by Lee and Seomun as "the capacity of a person to successfully fulfill the responsibilities expected from him within the norms of society". Nurses should not only have the care that meets the physical needs, but also have the adequacy of the skills that meet the psychosocial needs. Moral sensitivity has an important place in this holistic care provided by nurses.

Moral sensitivity is seeing the existence of ethical problems. It is also defined as the personal capacity to identify ethical problems in specific events in the relationship between patients and nurses. A nurse who does not have compassion for her patient cannot realize the situation of the patient and does not have moral sensitivity.

Generation Z, who will be in the nursing profession in the coming years, will have weak family ties, underdevelopment of their emotional intelligence, more narcissistic personalities, love to work independently, have high individuality and are less loyal than other generations. causes a low sense of compassion and therefore negatively affects their moral sensitivities. Since the Z generation is usually an only child and prevents socialization with people, their interpersonal relationships are weaker than other generations.

In this context, although there are studies in the literature stating that compassion has an important place in nursing education, no study has been found that examines the effect of compassion education on nursing students' compassion efficacy.

The aim of this thesis is to examine the effect of compassion education on compassion proficiency in nursing students.

ELIGIBILITY:
Inclusion Criteria:

* - voluntarily agree to participate in the research
* Continuing to work as an administrator in undergraduate places of Süleyman Demirel University
* Being able to understand and speak Turkish,
* No hearing and speech problems

Exclusion Criteria:

* Not voluntarily participating in the research
* Does not understand Turkish

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
The aim of this study is to examine the effect of compassion training on compassion proficiency in nursing students. | 6 weeks
  It will be collected from nursing students who volunteered to participate in the research by using the Compassion Adequacy Scale
The aim of this study is to examine the effect of compassion training on compassion | 6 weeks
  It will be collected from nursing students who volunteered to participate in the research by using the Modified Moral Sensitivity Scale for Nursing Students".

CONTACTS AND LOCATIONS:
Locations (1):
- Süleyman Demirel Üniversitesi, Isparta, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided